CLINICAL TRIAL: NCT05847088
Title: Intravitreal Dexamethasone Implant for Refractory Diabetic Macular Edema: Anatomical and Functional Outcomes of Treatment and Retreatment
Brief Title: Intravitreal Dexamethasone Implant for Refractory Diabetic Macular Edema:
Status: Completed | Type: Observational
Sponsor: Dar El Oyoun Hospital (Other)
Responsible Party: Principal Investigator, Wael Ahmed Ewais, Associate professor of Ophthalmology Cairo university, Dar El Oyoun Hospital
Other Study IDs: N-21-2023
Record Dates: First submitted 2023-04-05; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Calcium Dobesilate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Intravitreal Dexamethasone Implant for refractory Diabetic macular edema: — Intravitreal Dexamethasone implants (DEX) (0.7 mg) (Ozurdex, Allergan, Inc, Irvine, CA, USA) had been used with greater efficacy and safety in DME.
  Other Names: Ozurdex

SUMMARY:
We have been using DEX for refractory DME for a long time (since 2016). Thus, we are sharing our results , evaluating both anatomical and functional outcomes of DEX therapy for refractory DME.

DETAILED DESCRIPTION:
Our study aims at evaluating both anatomical and functional outcomes of DEX therapy for cases of refractory DME, with both a single injection, and /or with retreatments.

ELIGIBILITY:
Inclusion Criteria:

* • Age: 16 or older (Adults)

  * Sex: both
  * NTDME with CMT >300 u
  * < 10% reduction in CMT (than previous treatment)
  * < 50 u reduction in CMT (than previous treatment)
  * Worsening of BCVA > 1 line on E chart.
  * Duration since Previous treatment is: 3 months with DEX, 1 month with Anti-VEGF
  * Pseudophakic eyes
  * NPDR , PRP-treated PDR

Exclusion Criteria:

* • Phakic eyes

  * Uncontrolled Glaucoma (IOP > 24 mmHg, or cup disc ratio 0.8 or more)
  * Herpetic viral infection.
  * Untreated PDR

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Retrospective Review of records of patients with Non-tractional diffuse diabetic macular edema (NTDME), for whom Ozurdex had been used , in the period between 2016 and 2022.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Change in Central macular thickness (in microns) (CMT change ) | between baseline and 6 months
  Change in Central macular thickness (in microns) (CMT change )
Change in Best corrected visual acuity (BCVA change) ) | between baseline and 6 months
  lines of Change in Best corrected visual acuity (BCVA change) )

SECONDARY OUTCOMES:
Number of DEX injections | between baseline and 6 months
  Number of DEX injections
Shift to anti-VEGF during follow-up | between baseline and 6 months
  Shift to anti-VEGF during follow-up (Yes or No)
Duration of follow-up ( months) | between baseline and 6 months
  Duration of follow-up ( months)
CMT change > 100 u | between baseline and 6 months
  CMT change > 100 u (yes / No)
CMT change > 200 u | between baseline and 6 months
  CMT change > 200 u (yes / No)
BCVA change >= 2 lines | between baseline and 6 months
  BCVA change >= 2 lines (yes / No)
Complications : ocular hypertension, pseudo uveitis, endophthalmitis, RD | between baseline and 6 months
  Complications : ocular hypertension, pseudo uveitis, endophthalmitis, RD (yes / No)

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr alainy faculty of medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No